CLINICAL TRIAL: NCT00161122
Title: Effectiveness and Costs of Combined Influenza and Pneumococcal Vaccination in Pre-School Children With Recurrent Respiratory Tract Infections (RTI): a General Practice-Based Randomized Controlled Trial
Brief Title: Prevention of Respiratory Infections and MAnagement Among Children (PRIMAKid)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Primakid 1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2005-07

CONDITIONS: Recurrent Upper and Lower Respiratory Tract Infections (RTIs)

INTERVENTIONS:
Biological: trivalent inactivated influenza vaccine
Biological: combined heptavalent pneumococcal conjugate vaccine and trivalent inactivated influenza vaccine

SUMMARY:
The PRIMAKid trial is a general practice based double-blind randomized placebo-controlled trial on the effectiveness and costs of combined influenza and pneumococcal vaccination in pre-school children with recurrent respiratory tract infections. A target number of 660 children aged 18-72 months with a history of two or more general practitioner attended episodes of RTI, are included. Exclusion criteria are diseases accompanied by a high risk of recurrent RTI and conditions chronically treated with corticosteroids. Over a period of 7 to 22 months follow-up, the number of febrile RTI-episodes as primary outcome is assessed, and as secondary outcomes the severity and length of febrile RTI-episodes, medical visits / interventions, health-related quality of life and productivity loss of parents.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-72 months
* A history of two or more episodes of general practitioner attended RTIs

Exclusion Criteria:

* No intention to move within 12 months to another region
* Provision of informed consent
* Good mastering of the Dutch language
* Absence of chronic diseases such as asthma treated with corticosteroids or high-risk disease (such as palatoschisis, Down syndrome, cystic fibrosis, etc.)
* No previous influenza vaccination or pneumococcal vaccination or Hepatitis B vaccination
* No hypersensitivity to eggs and/or antibiotics, and/or serious history of serious adverse events through vaccination

Ages: 18 Months to 72 Months | Sex: All
Age Groups: Child
Enrollment: 660
Dates: Start 2003-09; Study Completion 2006-06

PRIMARY OUTCOMES:
number of febrile RTI-episodes

SECONDARY OUTCOMES:
severity and length of febrile RTI-episodes as well as medical consumption

CONTACTS AND LOCATIONS:
Overall Officials: Eelko Hak, PhD, Principal Investigator — Julius Center for Health Sciences and Primary Care, University Medical Center Utrecht
Locations (1):
- Julius Center for Health Sciences and Primary Care, University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Schonbeck Y, Sanders EA, Hoes AW, Schilder AG, Verheij TJ, Hak E. Rationale and design of the prevention of respiratory infections and management in children (PRIMAKid) study: a randomized controlled trial on the effectiveness and costs of combined influenza and pneumococcal vaccination in pre-school children with recurrent respiratory tract infections. Vaccine. 2005 Sep 30;23(41):4906-14. doi: 10.1016/j.vaccine.2005.05.021. PMID 16005552